CLINICAL TRIAL: NCT01703962
Title: Non Invasive IDentification of Gliomas With IDH1 Mutation by Free Plasmatic DNA Analysis, 2-hydroxyglutarate Dosage in the Urines and 2-hydroxyglutarate Detection by Brain SPEctro-MRI: Diagnostic and Follow-up Application (IDASPE)
Brief Title: Non Invasive IDentification of Gliomas With IDH1 Mutation
Acronym: IDASPE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-28; 2011-A01356-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Non Invasive Diagnosis of Glioma
Keywords: Glioma; IDH1; Spectroscopy; Plasma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples containing free DNA fragments Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with IDH1 R132H or wild type IDH1/IDH2 glioma

SUMMARY:
The recurrent mutation IDH1Arg132His leads to the cellular accumulation of D-2-hydroxyglutarate (2-HG), thus representing a diagnostic marker (this change is almost specific for gliomas) and prognostic (mutated gliomas have longer survival) of interest.

The main objective is to identify the patients with IDH1 mutated glioma by three complementary approaches -genetic (identification of IDH1 mutation in plasmatic DNA), biochemical (2-HG dosage in the urine of patients) and radiological (2-HG

DETAILED DESCRIPTION:
Our preliminary results indicate an extremely high amount of D-2HG in gliomas and CSF of the patients, and therefore the possibility to detect its presence by spectro-MRI, and to establish a non-invasive diagnosis of glioma with IDH1 mutation. Our goal is to identify and quantify by high-field MRI spectroscopy the presence of D-2HG to identify gliomas with IDH1 mutation. In parallel, we developed a technique for selective amplification of the mutated form of IDH1 (COLD PCR): by combining this technique with digital PCR, we already are able to detect IDH1 mutation from free plasma DNA with a sensitivity of 58% and a specificity of 100%. At the same time we have shown that D-2HG levels in urine of patients correlate with the status of the tumor IDH1.

The main objective is to identify using this triple approach (detection of the mutation on plasma DNA detection, detection of urinary D-2HG, detection of tumor D-2HG by spectro-MRI) patients with IDH1arg132His mutation, the secondary objective is to evaluate the value of these markers for patients follow-up and for differentiating recurrence from treatment induced damage. 40 patients with grade II and grade III gliomas (20 mutated, 20 non mutated) will be included and followed up for one year (five measurements are planned).

The first interest is diagnostic: the presence of the IDH1Arg132His mutation allows the diagnosis of glioma. This information is particularly valuable in patients not amenable to biopsy, because of the location of the tumor considered at risk, the general condition of the patient or the co-morbidities and medications. We hope also with these parameters to better monitor patient's follow-up, and to have a new method to differentiate tumor recurrence and radionecrosis or post-radiation leukoencephalopathy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* Affiliated to Health Insurance regimen (sécurité sociale)
* Patient of 18 years or more
* written informed consent
* Glioma grade II or III histologically proven
* Frozen samples available
* Known status IDH1/IDH2
* Presence of a measurable residual tumor (> 2 cm in diameter FLAIR)
* Karnofsky Performance Status (KPS)> 60

Exclusion Criteria:

* Contraindication to MRI *
* The rare patients with IDH2 mutation or with non Arg132His IDH1 mutation will be excluded
* Inability to provide informed consent
* Patient under guardianship or deprived of liberty by court

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the active file of patients with glioma II or III, followed at the Pitié-Salpetrière Hospital, and whose status is known for IDH1.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-03-14 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc SANSON, MDPhD, Principal Investigator — University of Pittsburgh
Locations (1):
- GH Pitié-Salpêtrière, 47 Bd de l'Hopital,, Paris, Sélectionner..., France

REFERENCES:
- [Derived] Branzoli F, Liserre R, Deelchand DK, Poliani PL, Bielle F, Nichelli L, Sanson M, Lehericy S, Marjanska M. Neurochemical Differences between 1p/19q Codeleted and Noncodeleted IDH-mutant Gliomas by in Vivo MR Spectroscopy. Radiology. 2023 Sep;308(3):e223255. doi: 10.1148/radiol.223255. PMID 37668523